CLINICAL TRIAL: NCT00948649
Title: Validation of a Novel Paradigm for Screening Medications for Nicotine Dependence
Brief Title: Effects of Chantix on Relapse Prevention for Smoking Cessation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Caryn Lerman, Ph.D., University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Screening
Other Study IDs: 805394
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2009-07

CONDITIONS: Nicotine Dependence
Keywords: Varenicline, Working memory
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Varenicline (Active Comparator): Participants will complete a 21-day study phase that will include a 10-day drug run-up and monitoring phase (days 1-10), a 3-day abstinence phase (days 11-13), and a programmed lapse (day 14) followed by a 7-day observation phase in which participants are asked to remain abstinent and will receive modest monetary reinforcement for doing so (days 15-21).
  Interventions: Drug: Varenicline
- Placebo (Placebo Comparator): Participants will complete a 21-day study phase that will include a 10-day drug run-up and monitoring phase (days 1-10), a 3-day abstinence phase (days 11-13), and a programmed lapse (day 14) followed by a 7-day observation phase in which participants are asked to remain abstinent and will receive modest monetary reinforcement for doing so (days 15-21).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Participants will take placebo pills for 21-days using the same regimen as the varenicline study period.
  Arms: Placebo
Drug: Varenicline — Day 1 - Day 3 0.5mg once daily Day 4 - Day 7 0.5mg twice daily Day 8 - End of Treatment 1.0mg twice daily
  Other Names: Chantix
  Arms: Varenicline

SUMMARY:
The goal of the proposed study is to validate an experimental paradigm to assess medication effects on smoking relapse following a brief (3-day) monitored period of smoking abstinence and a programmed cigarette lapse.

DETAILED DESCRIPTION:
The proposed human experiment will test the validity of a novel paradigm that may provide a method for distinguishing compounds that are likely to have efficacy from those that are not, before they are tested in more costly large-scale clinical trials. Specifically, in a within-subject (cross-over) behavioral pharmacology investigation of 60 smokers, we will test the effects of varenicline versus placebo on smoking behavior in the natural environment following a 3-day period of monitored abstinence and a programmed cigarette lapse. A positive signal for varenicline effects in this study would provide support for the sensitivity of the paradigm. In addition, following completion of all assessments, participants will be followed in a 13-week open-label varenicline smoking cessation trial to determine whether response to varenicline in the laboratory study predicts clinical response in the open-label trial.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will be 68 (34 male and 34 female) smokers aged 18-65, who smoke ≥ 10 cigarettes per day, provide a baseline CO reading ≥ 10 ppm and who plan to live in the area for the next 6-months.

Exclusion Criteria:

* Smoking Behavior

  1. Use of chewing tobacco or snuff
  2. Current enrollment or plans to enroll in another smoking cessation program in the next 5 months
  3. Plan to use other nicotine substitutes or smoking cessation treatments in the next 5 months
  4. Provide a baseline CO reading < 10 ppm

Alcohol/Drug Exclusion Criteria

1. History of substance abuse and/or currently receiving treatment for substance abuse (e.g., alcohol, opioids, cocaine, marijuana, or stimulants)
2. Current alcohol consumption that exceeds >25 standard drinks/week

Medication Exclusion Criteria

1. Current use or recent discontinuation (within last 14-days) of the following medications:

1. Any form of smoking cessation medication (zyban, wellbutrin, wellbutrin SR, Chantix, NRT)
2. Any form of anti-psychotic medications that includes:

   * antipsychotics,
   * atypical antipsychotics,
   * mood-stabilizers,
   * anti-depressants (tricyclics, SSRI's, MAOI's),
   * anti-panic agents,
   * anti-obsessive agents,
   * anti-anxiety agents, and
   * stimulants (e.g., Provigil, Ritalin).
3. Medication for chronic pain
4. Anti-coagulants
5. Any heart medications
6. Daily medication for asthma

Medical Exclusion Criteria

1. Women who are pregnant, planning a pregnancy, or lactating.
2. History or current diagnosis of psychosis, major depression or bipolar disorder, schizophrenia, or any Axis 1 disorder as identified by the SCID.
3. Serious or unstable disease within the past 6 months (e.g., cancer [except melanoma], heart disease, HIV).
4. History of epilepsy or a seizure disorder.
5. History or current diagnosis (last 6-months) of abnormal rhythms and/or tachycardia (>100 beats/minute); history or current diagnosis of COPD, cardiovascular disease (stroke, angina, coronary heart disease), heart attack in the last 6 months, uncontrolled hypertension (SBP>150 or DBP>90)
6. History of Kidney and/or liver failure (including transplant).
7. Wears a device to aid in hearing (hearing aid, cochlear implant, etc.).
8. Hearing threshold < 40 dB SPL at 1000 Hz.
9. Color blindness.

General Exclusion

1. Any medical condition or concomitant medication that could compromise participant safety or treatment, as determined by the Principal Investigator and/or Study Physician.
2. Inability to provide informed consent or complete any of the study tasks as determined by the Principal Investigator and/or Study Physician.
3. Any physical or visual impairment that may prevent the individual from using a computer keyboard or completing any study tasks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2006-09; Primary Completion 2007-08 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Days of abstinence following the programmed lapse | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Caryn Lerman, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Tobacco Use Research Center, University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Patterson F, Jepson C, Strasser AA, Loughead J, Perkins KA, Gur RC, Frey JM, Siegel S, Lerman C. Varenicline improves mood and cognition during smoking abstinence. Biol Psychiatry. 2009 Jan 15;65(2):144-9. doi: 10.1016/j.biopsych.2008.08.028. Epub 2008 Oct 8. PMID 18842256
- [Result] Rudnick ND, Strasser AA, Phillips JM, Jepson C, Patterson F, Frey JM, Turetsky BI, Lerman C, Siegel SJ. Mouse model predicts effects of smoking and varenicline on event-related potentials in humans. Nicotine Tob Res. 2010 Jun;12(6):589-97. doi: 10.1093/ntr/ntq049. Epub 2010 Apr 15. PMID 20395358
- [Result] Patterson F, Jepson C, Loughead J, Perkins K, Strasser AA, Siegel S, Frey J, Gur R, Lerman C. Working memory deficits predict short-term smoking resumption following brief abstinence. Drug Alcohol Depend. 2010 Jan 1;106(1):61-4. doi: 10.1016/j.drugalcdep.2009.07.020. Epub 2009 Sep 5. PMID 19733449
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273